CLINICAL TRIAL: NCT07098260
Title: DECIDE to Improve Maternal Mental Health Care Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Christina Kang-Yi, PhD, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro2024002663
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Mental Health Disorders

STUDY DESIGN:
Intervention Model Description: The DECIDE for MOM Provider Training will be adapted based on the DECIDE Provider Training model.10 Participants will take an asynchronous online DECIDE for MOM Provider Training (approximately 2 hours). DECIDE stands for Decide the problem; Explore the questions; Closed or open-ended questions; Identify the who, why, or how of the problem; Direct questions to your health care professional; Enjoy a shared solution. The 5 modules will cover shared decision-making, perspective-taking, patient activation, attributional errors, and being a responsive provider to perinatal individuals and include clinical illustrations developed for shared decision making in perinatal mental health care delivery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Providers (Experimental): The intervention targets nurses, midwives, primary care doctors, social workers, psychologists, case managers, counselors, peer specialists, and other obstetrics and gynecology care providers who provide perinatal health, mental health and or behavioral health care in hospitals or other healthcare organizations (e.g., home visit programs, State Medical Assistance and health services programs, Federally Qualified Health Centers). These providers receive an asynchronous online training that teaches them to communicate more effectively with their perinatal mental health care patients in order to improve shared decision making.
  Interventions: Behavioral: DECIDE for MOM Provider Training

INTERVENTIONS:
Behavioral: DECIDE for MOM Provider Training — Participants will take an asynchronous online DECIDE for MOM provider training (approximately 2 hours). DECIDE stands for Decide the problem; Explore the questions; Closed or open-ended questions; Identify the who, why, or how of the problem; Direct questions to your health care professional; Enjoy a shared solution. The 5 modules will cover shared decision-making, perspective-taking, patient activation, attributional errors, and being a responsive provider to perinatal individuals.

SUMMARY:
Appropriate training for perinatal mental health care is an important public health concern as mental health disorders are common pregnancy complications. Perinatal and mental health care providers report the difficulty of treating perinatal individuals due to insufficient information available regarding mental health treatment decisions, differences in beliefs and attitudes, and concerns about adverse effects on patients, such as self-harm and suicide. Effective shared decision-making skills can improve perinatal and mental health care providers' competencies to meet the unique decision needs of perinatal individuals, particularly those with mental health disorders. The proposed project titled "DECIDE to Improve Maternal Mental Health Care Delivery" aims to adapt the DECIDE Provider Training developed by Dr. Alegria and her team,1 to improve the rapid and wide dissemination and implementation of DECIDE in meeting the mental health needs of perinatal individuals. DECIDE stands for Decide the problem; Explore the questions; Closed or open-ended questions; Identify the who, why, or how of the problem; Direct questions to your health care professional; Enjoy a shared solution. The DECIDE provider training was developed based on theories of intergroup contact in social psychology and a patient-centered framework.28-30 DECIDE teaches mental health providers how to improve perspective-taking, reduce attributional errors, and increase receptivity to the client population.1,15-17 The proposed project will (1) make content adaptation (i.e., adding topical training content to fit perinatal mental health care) and process adaption (i.e., creating asynchronous training modules to reduce the burden for care providers) to the DECIDE Provider Training and (2) assess the acceptability, appropriateness, and usability of adapted DECIDE provider training for rapid and wide dissemination and implementation of DECIDE in maternal mental health care delivery.

DETAILED DESCRIPTION:
The project involves two phases. Phase 1: Adapt DECIDE to translate the knowledge of the DECIDE Provider Training into maternal mental health care. The investigators will use Iterative Decision-Making for the Evaluation of Adaptations (IDEA)20 and the Framework for Reporting Adaptations and Modifications-Enhanced (FRAME)21 as guiding frameworks for the adaptation. AHRQ's synthesis of research evidence for pharmacologic and nonpharmacologic treatments for maternal mental health care27 will be used as the guiding tool for selecting the key questions for shared decision making (SDM). The example questions include: whether to offer nonpharmacologic interventions alone or in combination with pharmacologic intervention for specific perinatal mental health conditions and which nonpharmacologic interventions for perinatal mental health lead to optimal patient outcomes. The core content of the DECIDE Provider Training will be retained in a 3-hour asynchronous training with 5 modules: shared decision-making, perspective-taking (understanding perinatal individuals' circumstances and perceptions), patient activation, attributional errors, and being a responsive provider to perinatal individuals. Vignettes will be created to address patient and provider concerns for perinatal mental health, such as pharmacological mental health treatment in relation to breastfeeding, pregnancy complications, maternal harms and child outcomes, patient sociodemographic factors, mental illness and prior pregnancy history, and patient preferences.

Stakeholder engagement to adapt DECIDE Provider Training: The investigators will establish a provider advisory board composed of perinatal and mental health care providers, and recruit 3 subject matter experts with expertise in perinatal mental health care, SDM, and health systems.

Recruitment of Provider Advisory Board: The investigators will recruit 5 provider advisory board members to guide adaptations to the DECIDE Provider Training. The members will include those who provide perinatal mental health care such as nurses, psychologists, social workers, midwives, counselors, peer specialists, and other providers. The advisory board will help identify content adaptations to be made to fit mental health treatment for perinatal individuals, review asynchronous training modules and vignettes, provide feedback on the provider training materials for revisions to be made, and advise how to best implement the adapted DECIDE provider training in health systems.

Recruitment of Subject Matter Experts: The investigators will recruit 3 subject matter experts with expertise in perinatal mental health, behavioral health, physical and emotional well-being, symptom management, and SDM. The experts will guide key content adaptations to be made to the provider training modules, provide relevant resources to create the content adaptation, co-develop scripts for the training vignettes with PI and Dr. Nakash (Consultant), and review provider training materials and make recommendations.

The investigators will conduct focus groups with the advisory board and subject matter experts to develop content adaptation and strategies for rapid and wide implementation of the DECIDE provider training in health systems. The focus groups will be held on the secure HIPPA-compliant Rutgers Zoom. Focus groups through Zoom have been reported to be an excellent method for programming and managing focus groups.39,40 A semi-structured topic guide consisting of broad, open-ended questions41 will include questions for structured stakeholder consultation/discussion on: (1) What are the anticipated key facilitators and barriers to using DECIDE as an SDM tool in health systems? (2) What are the components that must be included or avoided in the adaptations to the DECIDE Provider Training to ensure that perinatal and mental health providers in health systems use DECIDE skills taught?, and (3) What are appropriate and acceptable strategies to integrate the adapted DECIDE provider training into routine perinatal care processes?

Create, record, edit, and upload the adapted DECIDE provider training in Canvas: Gathering stakeholders' input, the investigators will develop training modules and scripts for vignettes, revise the training content and scripts through the iterative process of reviews and revisions by engaging the provider advisory board and the subject matter experts, and record training modules in Zoom webinars. Rutgers Online Education Services will produce video clips for vignettes based on the scripts provided, edit the video clips and recorded Zoom webinars, and upload them into Canvas.

Phase 2: Assess the acceptability, appropriateness, and usability of the adapted DECIDE provider training to build new knowledge of DECIDE implementation in perinatal mental health practice: The investigators will recruit 35 perinatal and mental health providers, including nurses, midwives, primary care doctors, social workers, psychologists, case managers, counselors, peer specialists, and other obstetrics and gynecology care providers who provide mental health care to perinatal individuals within health systems. Health systems include hospitals and other healthcare organizations (e.g., home visit programs, State Medical Assistance and health services programs, Federally Qualified Health Centers).

The participants will take the adapted DECIDE provider training: To identify the acceptability, appropriateness, and usability of asynchronous DECIDE provider training modules, the Acceptability, Feasibility, and Appropriateness Scale (AFAS)42 developed for the assessment of implementation outcomes for training in EBPs will be used. The measure demonstrates a good fit to the hypothesized three-factor structures (RMSEA = .058, CFI = .990, TLI = .987) and acceptable internal consistency (α = .86 to α = .91).42 The AFAS uses a 5-point Likert scale with 1 indicating "not at all" and 5 indicating "extremely." A few examples of the items are: "To what extent are you satisfied with the training you received and the practices covered?", "How comfortable are you with the practices contained within the training?", "How well do the information and practices fit with your overall approach to service delivery and the setting in which you provide care?" AFAS has demonstrated sensitivity to assessing workshop-specific perceptions about training acceptability and feasibility.42 The online assessment of acceptability, appropriateness, and usability will be conducted immediately after and one month after the training. Considering that immediately measuring acceptability, appropriateness, and usability can increase the correlation between appropriateness and usability but less highly correlated post-implementation of an intervention as providers perceive usability differently once they actually use the skills taught,44 providers who complete the training will be asked to also participate in the one-month follow-up evaluation.

Open-ended questions will be added to obtain detailed information on user acceptability, appropriateness and feasibility. The example questions include: (1) Share your experience of taking the asynchronous online training regarding login, course navigation, module organization, and other aspects of accessing the training (2) Did the training change how participants interact with perinatal individuals with mental health disorders? What are the specific examples? (3) What are the best strategies to effectively implement the DECIDE for MOM provider training within your organization?

The investigators will conduct focus groups with the training participants one month after the training to gain an in-depth understanding of participants' perceptions of acceptability, appropriateness, and usability of the adapted DECIDE provider training and thoughts about strategies to promote the high-quality implementation of the DECIDE training. The focus group meetings will be held on the secure HIPPA-compliant Rutgers Zoom. The semi-structured topic guide will be used for structured stakeholder consultation/discussion: (1) What are the key facilitators and barriers to practicing DECIDE skills taught in perinatal mental health care? (2) What are the components that must be included or avoided in the DECIDE provider training to ensure that mental health providers in health systems use it as an SDM tool?, and (3) What are appropriate and acceptable strategies to implement the DECIDE provider training as part of the routine perinatal mental health care at participants' organization?

ELIGIBILITY:
Inclusion Criteria:

* Perinatal or mental health care providers who currently provide perinatal mental health care within health systems
* Ages between 18 and 64
* Must be able to understand the training content in English and comfortably complete the assessments and share feedback in English

Exclusion Criteria:

* Healthcare providers who do not practice as part of a healthcare system
* Healthcare providers who do not practice in the U.S.
* Healthcare providers who do not currently provide perinatal mental health care

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability, Feasibility, and Appropriateness Scale (AFAS) | Immediately after and 1 month after the training
  The Acceptability, Feasibility, and Appropriateness Scale (AFAS)42 developed for the assessment of implementation outcomes for training in EBPs will be used. The measure demonstrates a good fit to the hypothesized three-factor structures (RMSEA = .058, CFI = .990, TLI = .987) and acceptable internal consistency (α = .86 to α = .91).42 The AFAS uses a 5-point Likert scale with 1 indicating "not at all" and 5 indicating "extremely." A few examples of the times are: "To what extent are you satisfied with the training you received and the practices covered?", "How comfortable are you with the practices contained within the training?", "How well do the information and practices fit with your overall approach to service delivery and the setting in which you provide care?" AFAS has demonstrated sensitivity to assessing workshop-specific perceptions about training acceptability and feasibility.42
Training Experience | Immediately after the training
  We will ask a set of open-ended questions to obtain detailed information on user acceptability, appropriateness and feasibility. The example questions include: (1) Share your experience of taking the asynchronous online training regarding login, course navigation, module organization, and other aspects of accessing the training (2) Did the training change how participants interact with perinatal individuals with mental health disorders? What are the specific examples? (3) What are the best strategies to effectively implement the DECIDE for MOM provider training within your organization?
Focus groups | 1 month after the training
  We will conduct focus groups with training participants one month after the training to gain an in-depth understanding of participants' perceptions of acceptability, appropriateness, and usability of adapted DECIDE and thoughts about strategies to promote the high-quality implementation of the DECIDE training.

CONTACTS AND LOCATIONS:
Overall Officials: Christina D Kang-Yi, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, the State University of New Jersey, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alegria M, Nakash O, Johnson K, Ault-Brutus A, Carson N, Fillbrunn M, Wang Y, Cheng A, Harris T, Polo A, Lincoln A, Freeman E, Bostdorf B, Rosenbaum M, Epelbaum C, LaRoche M, Okpokwasili-Johnson E, Carrasco M, Shrout PE. Effectiveness of the DECIDE Interventions on Shared Decision Making and Perceived Quality of Care in Behavioral Health With Multicultural Patients: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Apr 1;75(4):325-335. doi: 10.1001/jamapsychiatry.2017.4585. PMID 29466533